CLINICAL TRIAL: NCT02084069
Title: Atrovastatin for Preventing Atrial Fibrillation Following Open Cardiac Valve Repair
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Urmia University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: UMSU-Cardiology-2
Record Dates: First submitted 2014-03-08; First posted 2014-03-11 (Estimated); Results first posted 2015-02-04 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-02

CONDITIONS: Heart Valve Diseases
MeSH Terms: conditions — Heart Valve Diseases | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Treatment (Active Comparator): Atorvastatin 40 mg once daily from 3 days before surgery up to five days after surgery
  Interventions: Drug: Atorvastatin
- Control (Placebo Comparator): Placebo

INTERVENTIONS:
Drug: Atorvastatin
  Arms: Treatment

SUMMARY:
The purpose of the investigation is to determine whether Atrovastatin as anti-inflammatory agent can be effective in preventing from atrial fibrillation incidence in patients whom undergone open cardiac surgery for their heart valve repair.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 25 y/o
* No occurrence of intra- or post-operative cardiopulmonary arrest
* Not consuming drugs affecting atrial rhythm
* Having sinus rhythm before surgery
* Lack of paroxysmal atrial fibrillation history
* Only undergo heart valve surgery
* Lack of considerable heart ischemia needed atorvastatin use
* Routine cares in ward, post-operative ward, and intensive care unit were done

Exclusion Criteria:

* Lesser than 25 y/o
* History of atrial fibrillation
* History of taking anti-arrhythmic drugs
* History of implementing pacemakers
* Severe heart failure
* Renal failure
* Hepatic failure
* Severe pulmonary diseases
* Heart block or bradyarrhythmia
* Routine cares in ward, post-operative ward, and intensive care unit were not done
* Performing concomitant cardiac surgery except valve repair
* Having considerable heart ischemia needed atorvastatin use

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2013-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yousef Rezaei, M.D, Study Director — Seyyed-al-Shohada Heart Center, Urmia University of Medical Sciences
Locations (1):
- Seyyed-al-Shohada Heart Center, Urmia, West Azerbaijan Province, Iran

REFERENCES:
- [Derived] Dehghani MR, Kasianzadeh M, Rezaei Y, Sepehrvand N. Atorvastatin Reduces the Incidence of Postoperative Atrial Fibrillation in Statin-Naive Patients Undergoing Isolated Heart Valve Surgery: A Double-Blind, Placebo-Controlled Randomized Trial. J Cardiovasc Pharmacol Ther. 2015 Sep;20(5):465-72. doi: 10.1177/1074248414564869. Epub 2014 Dec 24. PMID 25540059
- See also: Related Info — http://umsu.ac.ir

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment | Control
Started | 29 | 29
Completed | 29 | 29
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled patients completed the study
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Control | Total
Number analyzed (Participants) | 29 | 29 | 58
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 54 [48 to 61] | 45 [39 to 52] | 49 [41 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 18 | 39
  Male | 8 | 11 | 19
Region of Enrollment [Number; unit: participants]
  Iran, Islamic Republic of | 29 | 29 | 58

OUTCOME MEASURES:

1. Primary Outcome: Atrial Fibrillation Incidence After Open Cardiac Valve Repair
Time Frame: Within 5 days after open cardiac valve repair
Measure: Number; unit: participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 29 | 29
participants | 6 | 13

ADVERSE EVENTS:
Arm/Group | Treatment | Control
Serious Adverse Events (participants affected / at risk) | 1/29 | 2/29
Other Adverse Events (participants affected / at risk) | 0/29 | 0/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=29) | Control (N=29)
Postoperative bleeding (Blood and lymphatic system disorders) | 1 (1) | 2 (2)

LIMITATIONS AND CAVEATS:
The sample size of this study was small

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No